CLINICAL TRIAL: NCT03252847
Title: An Open Label, Multi-centre, Phase I/II Dose Escalation Trial of a Recombinant Adeno-associated Virus Vector (AAV2/5-hRKp.RPGR) for Gene Therapy of Adults and Children With X-linked Retinitis Pigmentosa Owing to Defects in Retinitis Pigmentosa GTPase Regulator (RPGR)
Brief Title: Gene Therapy for X-linked Retinitis Pigmentosa (XLRP) - Retinitis Pigmentosa GTPase Regulator (RPGR)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MeiraGTx UK II Ltd (Industry)
Collaborators: Syne Qua Non Limited (Industry); Bionical Emas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MGT009
Record Dates: First submitted 2017-08-01; First posted 2017-08-17 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: X-Linked Retinitis Pigmentosa
Keywords: XLRP RPGR

STUDY DESIGN:
Intervention Model Description: Biological
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Part 1, Dose Escalation) (Experimental): Participants receive one of three doses of AAV5-RPGR
  Interventions: Genetic: AAV5-RPGR
- Phase 2 (Part 2; Expansion) (Experimental): Participants receive one of two doses of AAV5-RPGR
  Interventions: Genetic: AAV5-RPGR

INTERVENTIONS:
Genetic: AAV5-RPGR — Single, subretinal administration of AAV5-RPGR

SUMMARY:
Phase 1 of the study is a dose escalation of the subretinal administration of AAV5-hRKp.RPGR vector to assess the safety of this vector in participants with XLRP caused by mutations in RPGR. Participants enrolled in Phase 1 were assigned to a dose group based on when they enrolled (i.e., sequential assignment).

Phase 2 of the study is a cohort expansion of the subretinal administration of AAV5-hRKp.RPGR vector to assess the safety and efficacy of this vector in participants with XLRP caused by mutations in RPGR. Participants enrolled in Phase 2 were randomized to immediate or deferred treatment.

DETAILED DESCRIPTION:
This is an open-label phase 1/2 dose-escalation and cohort expansion trial to determine the safety and efficacy of subretinal administration of AAV5-hRKp.RPGR vector in participants with XLRP caused by mutations in RPGR.

ELIGIBILITY:
Key inclusion Criteria:

* Males aged 5 years or older
* Have X-linked retinitis pigmentosa confirmed by a retinal specialist (CI or PI)

Key exclusion Criteria:

• Have participated in another research study involving an investigational medicinal therapy for ocular disease within the last 6 months

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Bainbridge, Prof, Principal Investigator — University College, London
Locations (5):
- United States (3):
  - Massachusetts Eye and Ear Institute, Boston, Massachusetts
  - Kellogg Eye Center, Ann Arbor, Michigan
  - UPMC Eye Center, Pittsburgh, Pennsylvania
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Moorfields Eye Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michaelides M, Besirli CG, Yang Y, DE Guimaraes TAC, Wong SC, Huckfeldt RM, Comander JI, Sahel JA, Shah SM, Tee JJL, Kumaran N, Georgiadis A, Minnick P, Zeldin R, Naylor S, Xu J, Clark M, Anglade E, Wong P, Fleck PR, Fung A, Peluso C, Kalitzeos A, Georgiou M, Ripamonti C, Smith AJ, Ali RR, Forbes A, Bainbridge J. Phase 1/2 AAV5-hRKp.RPGR (Botaretigene Sparoparvovec) Gene Therapy: Safety and Efficacy in RPGR-Associated X-Linked Retinitis Pigmentosa. Am J Ophthalmol. 2024 Nov;267:122-134. doi: 10.1016/j.ajo.2024.05.034. Epub 2024 Jun 12. PMID 38871269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 sites (2 in the UK and 3 in the US) between 31 Jul 2017 and 18 Nov 2021. 49 participants were enrolled in the study; 4 participants discontinued before receiving treatment. The study consisted of 2 phases: dose escalation (Phase 1) followed by dose expansion (Phase 2). In Phase 1, 13 participants enrolled in 1 of 3 treatment groups. In Phase 2, 36 participants were randomized to an active treatment arm or a control arm with treatment deferred for 6 months.
Groups:
- Phase 1: Immediate Low Dose AAV5-hRKp.RPGR: Subretinal administration of a single low dose of AAV5-hRKp.RPGR in Phase 1 of the study.
  AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene.
- Phase 1: Immediate Intermediate Dose AAV5-hRKp.RPGR: Subretinal administration of a single intermediate dose of AAV5-hRKp.RPGR in Phase 1 of the study.
  AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene.
- Phase 1: Immediate High Dose AAV5-hRKp.RPGR: Subretinal administration of a single high dose of AAV5-hRKp.RPGR in Phase 1 of the study.
  AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene.
- Phase 2: Immediate Low Dose AAV5-hRKp.RPGR: Subretinal administration of a single low dose of AAV5-hRKp.RPGR in Phase 2 of the study.
  AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene.
- Phase 2: Immediate Intermediate Dose AAV5-hRKp.RPGR: Subretinal administration of a single intermediate dose of AAV5-hRKp.RPGR in Phase 2 of the study.
  AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene.
- Phase 2: Immediate High Dose AAV5-hRKp.RPGR: Subretinal administration of a single high dose of AAV5-hRKp.RPGR in Phase 2 of the study.
  AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene.
- Phase 2: Deferred Group: Treatment of participants in this Phase 2 study group was deferred for 6 months
Period: Overall Study
Arm/Group | Phase 1: Immediate Low Dose AAV5-hRKp.RPGR | Phase 1: Immediate Intermediate Dose AAV5-hRKp.RPGR | Phase 1: Immediate High Dose AAV5-hRKp.RPGR | Phase 2: Immediate Low Dose AAV5-hRKp.RPGR | Phase 2: Immediate Intermediate Dose AAV5-hRKp.RPGR | Phase 2: Immediate High Dose AAV5-hRKp.RPGR | Phase 2: Deferred Group
Started | 3 | 7 | 3 | 8 | 10 | 1 | 13
Completed | 3 | 7 | 2 | 8 | 9 | 1 | 13
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other: Patient decision | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Immediate Low Dose AAV5-hRKp.RPGR: Subretinal administration of a single low dose of AAV5-hRKp.RPGR in either Phase 1 or Phase 2 of the study (prespecified pooling).
  AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene
- Immediate Intermediate Dose AAV5-hRKp.RPGR: Subretinal administration of a single intermediate dose of AAV5-hRKp.RPGR in either Phase 1 or Phase 2 of the study (prespecified pooling).
  AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene
- Immediate High Dose AAV5-hRKp.RPGR: Subretinal administration of a single high dose of AAV5-hRKp.RPGR in either Phase 1 or Phase 2 of the study (prespecified pooling).
  AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene
- Deferred Group: Treatment of participants in this Phase 2 study group was deferred for 6 months
- Total: Total of all reporting groups
Arm/Group | Immediate Low Dose AAV5-hRKp.RPGR | Immediate Intermediate Dose AAV5-hRKp.RPGR | Immediate High Dose AAV5-hRKp.RPGR | Deferred Group | Total
Number analyzed (Participants) | 11 | 17 | 4 | 13 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 3 | 0 | 0 | 3
  Between 18 and 65 years | 11 | 14 | 4 | 13 | 42
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 11 | 17 | 4 | 13 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 11 | 16 | 4 | 11 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 10 | 15 | 3 | 13 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 1 | 5 | 14
  United Kingdom | 8 | 12 | 3 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting the Primary Outcome Defined as Any of the Below Events Occurring During the 9 Weeks Following Administration, at Least Possibly Related to the Advanced Therapy Investigational Medicinal Product (ATIMP), Not Surgery Alone.
Description: The primary outcome is defined as any of the below occurring during the 9 weeks following administration, at least possibly related to the Advanced Therapy Investigational Medicinal Product (ATIMP), not surgery alone:
  * Reduction in visual acuity by 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters or more
  * Severe unresponsive inflammation
  * Infective endophthalmitis
  * Ocular malignancy
  * Grade III or above non-ocular Suspected Unexpected Serious Adverse Reaction (SUSAR)
Time Frame: 9 weeks
Population: The primary endpoint was analyzed for participants in the dose escalation phase (i.e., study Phase 1) only
Measure: Count of Participants; unit: Participants
Groups:
- Immediate Low Dose AAV5-hRKp.RPGR: Subretinal administration of a single low dose of AAV5-hRKp.RPGR AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene
- Immediate Intermediate Dose AAV5-hRKp.RPGR: Subretinal administration of a single intermediate dose of AAV5-hRKp.RPGR AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene
- Immediate High Dose AAV5-hRKp.RPGR: Subretinal administration of a single high dose of AAV5-hRKp.RPGR AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene
- Deferred Group: Treatment of participants in this group was deferred for 6 months
Arm/Group | Immediate Low Dose AAV5-hRKp.RPGR | Immediate Intermediate Dose AAV5-hRKp.RPGR | Immediate High Dose AAV5-hRKp.RPGR | Deferred Group
Number analyzed (Participants) | 3 | 4 | 3 | 0
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Improvements in Visual Function as Assessed by Visual Acuity
Description: Change from baseline to Week 26 in best corrected visual acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) chart letter score. The direction of improvement from baseline is an increase in the number of ETDRS letters read over time.
Time Frame: Baseline and Month 6
Population: It was prespecified that the results of participants assigned to the low and intermediate dose groups in study Phase 1 and Phase 2 would be pooled and compared to the results of participants in the deferred group before treatment. Data were available for 25 participants in the Immediate Treatment Group and 13 participants in the Deferred Treatment Group
Measure: Mean (Standard Deviation); unit: Number of EDTRS letters
Groups:
- Immediate Treatment Group AAV5-hRKp.RPGR: Subretinal administration of a single dose of AAV5-hRKp.RPGR in adults AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene
Arm/Group | Immediate Treatment Group AAV5-hRKp.RPGR | Deferred Group
Number analyzed (Participants) | 25 | 13
Number of EDTRS letters | 0.6 (4.74) | -3.2 (3.87)

3. Secondary Outcome: Improvements in Retinal Function as Assessed by Static Perimetry
Description: The number of responders in point-by-point data in Static Perimetry within the full visual field over time.
  A responder at a single time point is defined as a participant with at least 5 of the same loci with ≥7 dB improvement from baseline at the specific time point and one time point prior.
Time Frame: Baseline and Month 6
Population: It was prespecified that the results of participants assigned to the low and intermediate dose groups in study Phase 1 and Phase 2 would be pooled and compared to the results of participants in the deferred group before treatment. Data were available for 23 participants in the Immediate Treatment Group and 10 participants in the Deferred Treatment Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Treatment Group AAV5-hRKp.RPGR | Deferred Group
Number analyzed (Participants) | 23 | 10
Participants | 6 | 2

4. Secondary Outcome: Quality of Life Measured by the Low Luminance Questionnaire (LLQ) Emotional Distress Domain Score
Description: Change from baseline to Week 26 in LLQ Emotional Distress Domain Score in adults. LLQ uses a scale from 0 to 100, with higher scores reflecting less impairment. A positive change from baseline reflects improvement, and a negative reflects worsening.
Time Frame: Baseline and Month 6
Population: It was prespecified that the results of participants assigned to the low and intermediate dose groups in study Phase 2 would be pooled and compared to the results of participants in the deferred group before treatment. Sixteen participants in the Immediate Treatment Group and all 9 participants in the Deferred Treatment Group completed the LLQ at baseline and Week 26.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Immediate Treatment Group AAV5-hRKp.RPGR | Deferred Group
Number analyzed (Participants) | 16 | 9
Units on a scale | 2.344 (20.1395) | -1.389 (8.7152)

5. Secondary Outcome: Quality of Life Measured by the Low Luminance Questionnaire (LLQ) Extreme Lighting Domain Score
Description: Change from baseline to Week 26 in LLQ Extreme Lighting Domain Score in adults. LLQ uses a scale from 0 to 100, with higher scores reflecting less impairment. A positive change from baseline reflects improvement, and a negative reflects worsening.
Time Frame: Baseline and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Immediate Treatment Group AAV5-hRKp.RPGR | Deferred Group
Number analyzed (Participants) | 16 | 9
Units on a scale | 2.956 (9.7080) | -8.059 (5.8453)

6. Secondary Outcome: Quality of Life Measured by the Low Luminance Questionnaire (LLQ) General Dim Lighting Domain Score
Description: Change from baseline to Week 26 in LLQ General Dim Lighting Domain score in adults. LLQ uses a scale from 0 to 100, with higher scores reflecting less impairment. A positive change from baseline reflects improvement, and a negative reflects worsening.
Time Frame: Baseline and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Immediate Treatment Group AAV5-hRKp.RPGR | Deferred Group
Number analyzed (Participants) | 16 | 9
Units on a scale | 4.115 (14.9706) | 1.852 (11.8056)

7. Secondary Outcome: Quality of Life Measured by the Low Luminance Questionnaire (LLQ) Mobility Domain Score
Description: Change from baseline to Week 26 in LLQ Mobility Domain Score in adults. LLQ uses a scale from 0 to 100, with higher scores reflecting less impairment. A positive change from baseline reflects improvement, and a negative reflects worsening.
Time Frame: Baseline and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Immediate Treatment Group AAV5-hRKp.RPGR | Deferred Group
Number analyzed (Participants) | 16 | 9
Units on a scale | 5.729 (15.8753) | 0.926 (6.5145)

8. Secondary Outcome: Quality of Life Measured by the Low Luminance Questionnaire (LLQ) Peripheral Vision Domain Score
Description: Change from baseline to Week 26 in LLQ Peripheral Vision Domain Score in adults. LLQ uses a scale from 0 to 100, with higher scores reflecting less impairment. A positive change from baseline reflects improvement, and a negative reflects worsening.
Time Frame: Baseline and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Immediate Treatment Group AAV5-hRKp.RPGR | Deferred Group
Number analyzed (Participants) | 16 | 9
Units on a scale | 1.563 (18.8116) | -1.852 (9.1076)

ADVERSE EVENTS:
Time Frame: Data are included from the signing of the ICF until the Month 12 visit.
Description: There were 3 SAEs (all non-fatal) reported during the study: 2 in the immediate treatment group (preferred terms retinal detachment and uveitis) and 1 in the deferred treatment group after surgery (preferred term intraocular pressure increased).
Groups:
- Deferred Group - Before Treatment (Control Group): Treatment of participants in this Phase 2 group was deferred for 6 months. Data from these deferred-treatment participants (i.e., the Control Group) are included from the signing of the ICF until the time of surgery
- Deferred Group - Low Dose AAV5-hRKp.RPGR - After Treatment: Subretinal administration of a single low dose of AAV5-hRKp.RPGR AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene. Treatment of participants in this Phase 2 group was deferred for 6 months. Data from these deferred treatment participants are included from the time of surgery until the end of the study.
- Deferred Group - Intermediate Dose AAV5-hRKp.RPGR - After Treatment: Subretinal administration of a single intermediate dose of AAV5-hRKp.RPGR AAV5-hRKp.RPGR: AAV gene therapy for defects in the RPGR gene.
  Treatment of participants in this Phase 2 group was deferred for 6 months. Data from these deferred treatment participants are included from the time of surgery until the end of the study.
Arm/Group | Immediate Low Dose AAV5-hRKp.RPGR | Immediate Intermediate Dose AAV5-hRKp.RPGR | Immediate High Dose AAV5-hRKp.RPGR | Deferred Group - Before Treatment (Control Group) | Deferred Group - Low Dose AAV5-hRKp.RPGR - After Treatment | Deferred Group - Intermediate Dose AAV5-hRKp.RPGR - After Treatment
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/17 | 0/4 | 0/13 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/17 | 0/4 | 0/13 | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 11/11 | 17/17 | 4/4 | 1/13 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Low Dose AAV5-hRKp.RPGR (N=11) | Immediate Intermediate Dose AAV5-hRKp.RPGR (N=17) | Immediate High Dose AAV5-hRKp.RPGR (N=4) | Deferred Group - Before Treatment (Control Group) (N=13) | Deferred Group - Low Dose AAV5-hRKp.RPGR - After Treatment (N=7) | Deferred Group - Intermediate Dose AAV5-hRKp.RPGR - After Treatment (N=6)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Assessed by the Investigator as ATIMP-related
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Assessed by the Investigator as ATIMP-related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Low Dose AAV5-hRKp.RPGR (N=11) | Immediate Intermediate Dose AAV5-hRKp.RPGR (N=17) | Immediate High Dose AAV5-hRKp.RPGR (N=4) | Deferred Group - Before Treatment (Control Group) (N=13) | Deferred Group - Low Dose AAV5-hRKp.RPGR - After Treatment (N=7) | Deferred Group - Intermediate Dose AAV5-hRKp.RPGR - After Treatment (N=6)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 5 | 9 | 2 | 0 | 4 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 1
Intraocular pressure decreased (Investigations) | 2 | 1 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 2 | 0 | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 8 | 11 | 4 | 0 | 2 | 3
Anterior chamber cell (Eye disorders) | 4 | 9 | 3 | 0 | 2 | 2
Visual acuity reduced (Eye disorders) | 6 | 8 | 2 | 0 | 6 | 6
Eye inflammation (Eye disorders) | 3 | 5 | 0 | 0 | 2 | 1
Foreign body sensation in eyes (Eye disorders) | 1 | 5 | 2 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 3 | 4 | 1 | 0 | 2 | 1
Cystoid macular oedema (Eye disorders) | 2 | 3 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 2 | 3 | 0 | 0 | 2 | 1
Conjunctival hyperaemia (Eye disorders) | 2 | 2 | 0 | 0 | 3 | 0
Posterior capsule opacification (Eye disorders) | 1 | 3 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 4 | 0 | 0 | 2 | 0
Uveitis (Eye disorders) | 0 | 2 | 2 | 0 | 0 | 0
Cataract (Eye disorders) | 2 | 0 | 1 | 0 | 0 | 0
Retinal cyst (Eye disorders) | 0 | 2 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 2 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 2 | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03252847/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT03252847/SAP_001.pdf